CLINICAL TRIAL: NCT04020432
Title: Knowledge Assessment of Pregnant or Childbearing Age Women About Pictograms Associated With the Danger of Certain Medicines Taken During Pregnancy.
Brief Title: Knowledge Assessment of Women About Pictograms Associated With the Danger of Medicines Taken During Pregnancy
Acronym: ECOFP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier HIRSON (Unknown)
Responsible Party: Sponsor
Other Study IDs: PI2018_843_0042
Record Dates: First submitted 2019-07-12; First posted 2019-07-16 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Knowledge, Attitudes, Practice; Pregnancy Related
Keywords: knowledge; medicine; pictogram; pregnant woman; childbearing age woman
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant women: Pregnant women are coming to their monthly consultation. A quantitative questionnaire has been created under primary and secondary assumptions. Questionnaires are going to be distributed to women who are agree to participate to this study. The questionnaires are going to be delivered by the investigators.
  Pregnant women can answer the questionnaire in the waiting room of consultation's services. The questionnaire will be anonymous and the return of questionnaires will be made personally.
  Interventions: Behavioral: questionary
- childbearing age women: Women of childbearing age, who are coming for a gynecological consultation. A quantitative questionnaire has been created under primary and secondary assumptions. Questionnaires are going to be distributed to women who are agree to participate to this study. The questionnaires are going to be delivered by the investigators.
  Childbearing age women can answer the questionnaire in the waiting room of consultation's services. The questionnaire will be anonymous and the return of questionnaires will be made personally.
  Interventions: Behavioral: questionary

INTERVENTIONS:
Behavioral: questionary — A quantitative questionnaire has been created under primary and secondary assumptions. Questionnaires are going to be distributed to women who are agree to participate to this study. The questionnaires are going to be delivered by the investigators.
  Women can answer the questionnaire in the waiting room of consultation's services. The questionnaire will be anonymous and the return of questionnaires will be made personally.

SUMMARY:
Women's awareness about the danger of certain medicines taken during pregnancy presents a real public health issue. To enhance awareness and information for women and healthcare professionals, new pictograms " pregnant women " appeared on medication boxes, on October 16, 2017. These new pictograms can change women's perception of self-medication during pregnancy and of the danger of taking certain medicines for the unborn development. Furthermore, the investigators can wonder if the meaning of these pictograms is well understood. Therefore, the study's primary aim is to assess the knowledge of pregnant or childbearing age women about the pictograms associated with the danger of certain medicines taken during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women who agree to participate to the study
* women who understand french language (oral and written)
* pregnant women and women of childbearing age from 18 to 45 years old.

Exclusion Criteria:

* Women who have already answered the questionnaire
* women who don't want to answer the questionnaire
* women who don't understand french language
* women who are under the age of 18 or over the age of 45

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — this study is includying only pregnant and childbearing age women
Study Population: pregnant or childbearing age women between 18 and 45 years old.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Medication pictogram women knowledge measure | day 0
  Determination of women knowledge about pictograms associated with the danger of certain medicines during pregnancy by analysing the questionnaire responses

SECONDARY OUTCOMES:
Medication pictogram women information measure | day 0
  Determination of women information about pictograms associated with the danger of certain medicines during pregnancy by analysing the questionnaire responses

CONTACTS AND LOCATIONS:
Overall Officials: Alice Rousseaux, Principal Investigator — CH Hirson
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No